CLINICAL TRIAL: NCT05472883
Title: Identification of Human Circulating Adipocyte and Muscle Biomarkers Potentially Predictive of Diabetes Remission After Bariatric Surgery in Obese and Type 2 Diabetic Subjects.
Brief Title: Identification of Human Biomarkers Predictive of Diabetes Remission in Type 2 Diabetes Patient (BARIAKINES)
Acronym: BARIAKINES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/21/0614
Record Dates: First submitted 2022-06-13; First posted 2022-07-25 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Obesity; Bariatric Surgery Candidate; Proteins; Biomarkers
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is an exploratory pilot study, comparing for the first time in humans, the remission of type 2 diabetes, one year after bariatric surgery, with regard to circulating concentrations of 9 candidate proteins measured at T0.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Experimental): This arm consists of obese patients with type 2 diabetes who are scheduled for bariatric surgery.
  Interventions: Procedure: blood samples; Procedure: collection of body tissues; Procedure: routine care procedure

INTERVENTIONS:
Procedure: blood samples — - Research blood sample: 2 additional tubes compared to the classic sample for the analysis of the 9 research molecules.
Procedure: collection of body tissues — removal of intra-abdominal fat and muscle tissue
Procedure: routine care procedure — * Routine care blood sample: Full vitamin panel, CBC, liver panel, urea, creatinine, blood ionogram, blood calcium, phosphorus, magnesium at all visits, except the morning of surgery when only ß HCG (for women of childbearing age), HbA1c.
  * clinical examination : weight, height, waist measurement, cardiovascular examination, digestive system examination.
  * dosage of ß HCG for womens.

SUMMARY:
This study focuses on identifying potentially predictive human circulating adipocyte and muscle biomarkers of diabetes remission after bariatric surgery in obese type 2 diabetic (T2D) subjects.

DETAILED DESCRIPTION:
The study team at the Institute of Metabolic and Cardiovascular Diseases has recently identified several potential biomarkers (secreted by skeletal muscle and adipose tissue) of glucose homeostasis control using secretomic and metabolomic analyses. The goal of this study is to assess whether the addition of 9 adipocytes and myocytes plasma level could be associated with type 2 diabetes remission one year after bariatric surgery and would improve established clinical models of prediction of diabetes remission.

Thus, obese type 2 diabetes patients undergoing bariatric surgery will have 2 blood samples, a muscle sample and one adipose tissue sample withdrawn during the study. From those samples, concentrations of 9 candidate proteins is measured : GDF6, INHBB, IL17B, TGFB2, TIMP1, VTN, MDK, GDF15, and apoM

ELIGIBILITY:
Inclusion Criteria:

* Obese patients of at least grade 2 (body mass index ≥ 35 kg/m²)
* Type 2 diabetics
* About to undergo bariatric surgery at the Toulouse University Hospital
* Affiliated or beneficiaries of a social security plan.
* Having provided a free, informed and written consent, signed

Exclusion Criteria:

* Type 1 diabetic subjects or Maturity-Onset Diabetes of the Youth.
* Pregnant and breastfeeding women.
* Vulnerable persons as defined in the Public Health Code: protected adults (guardianship, curators), unable to express their consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between plasma levels of 9 target molecules and diabetes remission | Immediately before the Surgery (day 0)
  The correlation between plasma levels of 9 target molecules (1 for each molecule) and diabetes remission will be evaluated through plasmatic dosages.
  The plasma determination of apolipoprotein M will be performed by mass spectrometry, and the 8 other molecules will be determined by the ELISA technique. The dosage is measured in mmol/l.
  Complete remission of T2DM will be defined according to the following criteria: HbA1c < 5.7% and fasting blood glucose < 5.6 mmol/l.
  Partial remission of T2DM will be defined as: HbA1c between 5.7 and 6.5% and fasting blood glucose between 5.6 and 6.9 mmol/l without any antidiabetic treatment. Finally, the absence of remission will include patients whose HbA1c is greater than or equal to 6.5% or fasting blood glucose greater than or equal to 7 mmol/l with one or more antidiabetic treatments.
Correlation between plasma levels of 9 target molecules and diabetes remission | At 3 months post-surgery
  The correlation between plasma levels of 9 target molecules (1 for each molecule) and diabetes remission will be evaluated will be evaluated through plasmatic dosages.
  The plasma determination of apolipoprotein M will be performed by mass spectrometry, and the 8 other molecules will be determined by the ELISA technique. The dosage is measured in mmol/l.
  Complete remission of T2DM will be defined according to the following criteria: HbA1c < 5.7% and fasting blood glucose < 5.6 mmol/l.
  Partial remission of T2DM will be defined as: HbA1c between 5.7 and 6.5% and fasting blood glucose between 5.6 and 6.9 mmol/l without any antidiabetic treatment. Finally, the absence of remission will include patients whose HbA1c is greater than or equal to 6.5% or fasting blood glucose greater than or equal to 7 mmol/l with one or more antidiabetic treatments.
Correlation between plasma levels of 9 target molecules and diabetes remission | At 12 months post-surgery
  The correlation between plasma levels of 9 target molecules (1 for each molecule) and diabetes remission will be evaluated will be evaluated through plasmatic dosages.
  The plasma determination of apolipoprotein M will be performed by mass spectrometry, and the 8 other molecules will be determined by the ELISA technique. The dosage is measured in mmol/l.
  Complete remission of T2DM will be defined according to the following criteria: HbA1c < 5.7% and fasting blood glucose < 5.6 mmol/l.
  Partial remission of T2DM will be defined as: HbA1c between 5.7 and 6.5% and fasting blood glucose between 5.6 and 6.9 mmol/l without any antidiabetic treatment. Finally, the absence of remission will include patients whose HbA1c is greater than or equal to 6.5% or fasting blood glucose greater than or equal to 7 mmol/l with one or more antidiabetic treatments.

SECONDARY OUTCOMES:
Areas under the ROC curves of different logistic regression models fitted to known clinical prediction scores (DiaRem, Ad-DiaRem). | At 3 months post-surgery
  The DiaRem and Ad-DiaRem scores are weighted scoring systems based on initial pre-surgical factors that were specifically created to predict remission of type 2 diabetes after bariatric surgery.
Areas under the ROC curves of different logistic regression models fitted to known clinical prediction scores (DiaRem, Ad-DiaRem). | At 12 months post-surgery
  The DiaRem and Ad-DiaRem scores are weighted scoring systems based on initial pre-surgical factors that were specifically created to predict remission of type 2 diabetes after bariatric surgery.
the kinetics of the plasma levels of each of the 9 molecules studied | Immediately before the Surgery (day 0)
  the kinetics of the plasma levels of each of the 9 molecules will be studied by measuring each factor on an empty stomach: the day of the operation in the digestive surgery department.
the kinetics of the plasma levels of each of the 9 molecules studied | At 3 months after the surgery
  the kinetics of the plasma levels of each of the 9 molecules will be studied by measuring each factor on an empty stomach: the day of the operation in the digestive surgery department.
the kinetics of the plasma levels of each of the 9 molecules studied | At 12 months after the surgery
  the kinetics of the plasma levels of each of the 9 molecules will be studied by measuring each factor on an empty stomach: the day of the operation in the digestive surgery department.
The expression level of genes encoding 9 biomarkers in the adipocyte and the muscle cell | At the day of the inclusion
  The expression level of the genes encoding 9 biomarkers in the adipocyte and the muscle cell will be evaluated by measuring the mRNA quantities of the genes of these 9 proteins
The expression level of genes encoding 9 biomarkers in the adipocyte and the muscle cell | At 3 months after surgery
  The expression level of the genes encoding 9 biomarkers in the adipocyte and the muscle cell will be evaluated by measuring the mRNA quantities of the genes of these 9 proteins
The expression level of genes encoding 9 biomarkers in the adipocyte and the muscle cell | At 12 months after surgery
  The expression level of the genes encoding 9 biomarkers in the adipocyte and the muscle cell will be evaluated by measuring the mRNA quantities of the genes of these 9 proteins

CONTACTS AND LOCATIONS:
Overall Officials: Emilie MONTASTIER, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, France